CLINICAL TRIAL: NCT04892641
Title: A Phase 1, Double-blind, Placebo-controlled, Dose-Ranging Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Food Effect of Epetraborole Tablets Administered for up to 28 Days in Healthy Adult Subjects
Brief Title: Phase 1 Study of Epetraborole Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AN2 Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: EBO-101
Record Dates: First submitted 2021-05-11; First posted 2021-05-19 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Epetraborole for Dose Ranging (Experimental): Epetraborole hydrochloride 250 mg, 500 mg, 750 mg, or 1000 mg PO q24h or 500 mg or 1000 mg PO q48h
  Interventions: Drug: Epetraborole
- Placebo for Dose Ranging (Placebo Comparator): Matching placebo for dose ranging
  Interventions: Drug: Placebo
- Epetraborole for Food Effect (Experimental): Food effect cohort, single dose in fed and fasted conditions, dosage to be determined based on pharmacokinetics data obtained from previous cohorts
  Interventions: Drug: Epetraborole
- Placebo for Food Effect (Placebo Comparator): Food effect cohort, single dose in fed and fasted conditions, dosage to be determined based on pharmacokinetics data obtained from previous cohorts
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Epetraborole — Epetraborole hydrochloride 250 mg tablets for oral administration
  Other Names: AN2-501971
  Arms: Epetraborole for Dose Ranging; Epetraborole for Food Effect
Drug: Placebo — Matching placebo for 250 mg epetraborole hydrochloride tablets for oral administration
  Arms: Placebo for Dose Ranging; Placebo for Food Effect

SUMMARY:
This is a Phase 1b double-blind, placebo-controlled, dose-ranging study to evaluate the safety, tolerability, PK, and food effect of epetraborole tablets administered to healthy adult subjects for up to 28 days.

DETAILED DESCRIPTION:
Up to 56 healthy male and female adult subjects will be enrolled into one of 7 Dose Cohorts (Dose Cohorts 1 to 7; n = 8 per cohort). Cohort 7 (n = 8) is a Food Effect Cohort and subjects will receive a single dose of epetraborole or placebo in a Fasted state (Period 1) followed by a second dose of the same Investigational Product (IP) in a Fed state (Period 2) after a washout period of at least 7 days (+3 days). The dose of IP to be administered in Cohort 7 will be determined based on the Safety Monitoring Group recommendation following evaluation of safety and available PK data (at least 14 days) in Cohort 1 through Cohort 6. Up to 16 additional subjects may be included for the purposes of cohort expansion or to explore a dose intermediate to previously evaluated doses.

Subjects in each Dose Cohort (n=8) will be randomized 3:1 to receive epetraborole (n=6) or matching placebo (n=2) and will receive oral doses of epetraborole or placebo. Investigational product will be administered with approximately 240 mL (8 fluid ounces) of non-carbonated water to each subject following an overnight fast of at least 8 hours, except for Period 2 (Fed) of Cohort 7. Subjects will be required to fast for a minimum of 2 hours following administration of IP.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all the following criteria will be considered for inclusion in the study:

1. Healthy adult males and/or females of 18 to 65 years of age (inclusive) at the time of Screening.
2. Willing and able to provide written informed consent.
3. Body mass index (BMI) ≥ 18.0 and ≤ 30.0 kg/m2 and weight between 40.0 kg and 100.0 kg (inclusive) at Screening.
4. Medically healthy without CS abnormalities at the Screening Visit or Day -1, including:

   1. Physical examination, vital signs including temperature, HR, respiratory rate, and blood pressure
   2. Triplicate ECGs taken at least 1 minute apart with QTcF interval duration ≤ 450 msec obtained as an average from the triplicate Screening and pre-dose Day 1 ECGs after at least 5 minutes in a semi-supine, quiet rest position
   3. Hematological parameters (including hemoglobin, hematocrit, red blood cells [RBC], packed cell volume [PCV], mean corpuscular volume [MCV], mean corpuscular hemoglobin [MCH], mean corpuscular hemoglobin concentration [MCHC], red cell distribution width [RDW], platelet count, white blood cell [WBC] and differential, and reticulocytes) are equal to or greater than the lower limit of normal (LLN) of the normal range of the reference laboratory
   4. Estimated creatinine clearance (CrCl) or glomerular filtration rate (GFR) < 80 mL/min using Cockcroft-Gault formula (calculated creatinine clearance or GFR = [{140-Age} × Weight {in kg}] \ [72 × Serum creatinine {in mg/dL}] × 0.85 [if female]); ALT and AST equal to or ≤ 1.5 times the ULN; results of all other clinical chemistry and urine analytes without any CS abnormality Note: Discussion between the PI and the Sponsor Medical Monitor (MM) is required regarding any potentially CS abnormal laboratory value during the pre-dose period.
5. Non-smoker (including tobacco, e-cigarettes, nicotine patches or marijuana) for at least 1 month prior to randomization, which will be confirmed by urine cotinine test at Screening and on Day -1 (admission).
6. Willing and able to comply with all study assessments and adhere to the protocol schedule, including the entire confinement period and the F/U visits.
7. Have suitable venous access for blood sampling.
8. Women of childbearing potential (WOCBP) must have a negative pregnancy test at Screening and on Day -1 (admission) and be willing to have additional pregnancy tests, as required, throughout the study.

   WOCBP must agree to and comply with using 1 barrier method (e.g., female condom or male partner using a condom) plus 1 other highly effective method of birth control (e.g., oral contraceptive pills [OCPs], long-acting implantable hormones, injectable hormones, intrauterine device [IUD], vasectomized partner), or sexual abstinence, for the duration of the study (from signing of consent to final F/U visit) and for 30 days after last IP administration.

   WOCBP must also agree not to donate ova or oocytes (i.e., human eggs) during the study, and for one menstrual cycle after completion of the study To be considered of non-childbearing potential, a female must have either a tubal ligation, hysterectomy, bilateral salpingo-oophrectomy, or menopause (last menstruation > 12 months and follicle-stimulating hormone [FSH] levels ≥ 40 IU/mL at Screening); provision of written documentation is not required for female sterilization and oral confirmation is adequate.

   Female subjects who are in same-sex relationships are not required to use contraception.
9. Males must be surgically sterile (> 30 days since vasectomy), abstinent, or if engaged in sexual relations with a WOCBP, the subject and his partner must be surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or using an acceptable, highly effective contraceptive method from Screening until study completion, including the F/U period. Acceptable methods of contraception include the use of condoms and the use of an effective contraceptive for the female partner that includes: OCPs, long-acting implantable hormones, injectable hormones, a vaginal ring or an IUD. Subjects with same-sex partners are eligible when this is their preferred and usual lifestyle.

   Males must not donate sperm for the duration of the study (from signing of consent to final F/U visit) and for 90 days after last IP administration.
10. Subjects must agree to adhere to the current state and national advice regarding minimizing exposure to coronavirus disease of 2019 (COVID-19) from the first Screening Visit until the final F/U visit.

Exclusion Criteria:

1. Pregnant or lactating at Screening or planning to become pregnant (self or partner) at any time during the study, including the F/U period.
2. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic or neurological disease, including any acute illness or major surgery within the past 3 months determined by the PI to be CS.
3. Iron, B12 or folate outside of the normal range at Screening and any history of anemia (e.g. iron deficiency, B12 or folate deficiency, or hemoglobinopathy).
4. Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years prior to Screening.
5. Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome).
6. Has/had febrile illness or symptomatic viral, bacterial (including upper respiratory tract infection) or fungal infection within 2 weeks prior to randomization.
7. Unable to swallow solid, oral dosage forms whole with the aid of water.
8. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) antibody.
9. Positive urine drug screen or alcohol breath test at Screening or Day -1, or history of substance abuse or alcohol abuse (defined as greater than 2 standard drinks on average each and every day, where 1 standard drink is defined as containing 10 g of alcohol and is equivalent to 1 can or stubby of mid-strength beer, 30 mL nip of spirits, or 100 mL of wine) within the previous 6 months.
10. Use of any prescription medication or any over the counter (OTC) medication, including erythropoietin stimulating agents, herbal products and vitamins, within 7 days prior to randomization.

    Note: An exception is made for hormonal contraceptives and intermittent, as-needed acetaminophen or nonsteroidal anti-inflammatory drugs (NSAIDs) for the treatment of transient headache or any other minor ache/pain. Discussion between the PI and the Sponsor MM is encouraged regarding the acceptability of the prior use of any medications during the pre-dose period.
11. Any vaccinations or planned vaccinations (including COVID-19 and influenza) within 14 days prior to dosing on Day 1 and for the duration of the study (up to the F/U visit).
12. Documented significant hypersensitivity reaction or anaphylaxis to any medication, which in the opinion of the Investigator could compromise subject safety.
13. Donation of blood or plasma within 30 days prior to randomization, or loss of whole blood of more than 500 mL within 30 days prior to randomization, or past receipt of a blood transfusion at any time.
14. Received an investigational intervention (including an investigational vaccine) or used an invasive investigational medical device within 30 days (or 5 half-lives whichever is longer) prior to Day 1.
15. Any other condition or prior therapy, which, in the opinion of the PI, would make the volunteer unsuitable for this study, including unable to cooperate fully with the requirements of the study protocol or likely to be non-compliant with any study requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-02-26 (Actual); Study Completion 2022-02-26 (Actual)

PRIMARY OUTCOMES:
Evaluate the Incidence of Treatment Emergent Adverse Events at Baseline and Through Study Completion | From Day 1 through last follow-up visit (7 days after last dose)
  Incidence, relatedness, and severity of adverse events
Evaluate Physical Examination Abnormalities from Baseline Through Study Completion | From Day 1 through last follow-up visit (7 days after last dose)
  Incidence of physical exam abnormalities
Evaluate Change in Vital Signs from Baseline Through Study Completion | From Day 1 to follow-up visit through last follow-up visit (7 days after last dose)
  Incidence of changes in blood pressure, pulse, respiratory rate, and temperature
Evaluate Changes in 12-lead ECG Measurements from Baseline Through Study Completion | From Day 1 to follow-up visit through last follow-up visit (7 days after last dose)
  Incidence of changes in 12-lead ECG parameters from baseline
Evaluate Changes in Clinical Laboratory Tests from Baseline Through Study Completion | From Day 1 to follow-up visit through last follow-up visit (7 days after last dose)
  Incidence of changes in clinical laboratory measurements from baseline
Characterize the PK Profile of Epetraborole: Maximum Plasma Concentration | From Day 1 to follow-up visit through last follow-up visit (7 days after last dose)
  Determination of the maximum plasma concentration (Cmax)
Characterize the PK Profile of Epetraborole: Minimum Steady State Plasma Concentration During a Dosage Interval | From Day 1 to follow-up visit through last follow-up visit (7 days after last dose)
  Determination of the minimum steady state plasma drug concentration during a dosage interval (Cmin)
Characterize the PK Profile of Epetraborole: Time to Maximum Plasma Concentration | From Day 1 to follow-up visit through last follow-up visit (7 days after last dose)
  Determination the time to maximum plasma concentration (Tmax)
Characterize the PK Profile of Epetraborole: Area Under the Plasma Concentration Versus Time Curve from Time 0 to the Last Time Point Evaluated | From Day 1 to follow-up visit through last follow-up visit (7 days after last dose)
  Determine the area under the plasma concentration versus time curve from time 0 to the last time point evaluated (AUC0-t) with the plasma concentration at time "t" being the last measurable concentration
Characterize the PK Profile of Epetraborole: Area Under the Plasma Concentration Versus Time Curve from Time 0 to Infinity | From Day 1 to follow-up visit through last follow-up visit (7 days after last dose)
  Determine area under the drug concentration versus time curve, from time zero to infinity (AUC0-inf)
Characterize the PK Profile of Epetraborole: Last Quantifiable Concentration | From Day 1 to follow-up visit through last follow-up visit (7 days after last dose)
  Determine the actual time of last quantifiable concentration used in the determination of AUC0-last (Tlast)
Characterize the PK Profile of Epetraborole: Terminal Half-Life | From Day 1 to follow-up visit through last follow-up visit (7 days after last dose)
  Determine the apparent terminal half-life (t½)
Characterize the PK Profile of Epetraborole: Terminal Elimination Rate Constant | From Day 1 to follow-up visit through last follow-up visit (7 days after last dose)
  Determine apparent terminal elimination rate constant (Kel)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Molga, M.D., Principal Investigator — CMAX Clinical Research
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No